CLINICAL TRIAL: NCT05188274
Title: A Multicenter, Randomized, Double-blind, and Placebo-controlled Clinical Study to Evaluate the Safety and Efficacy of T92 in Pediatric Patients With Tourette Syndrome
Brief Title: A Clinical Study to Evaluate the Safety and Efficacy of T92 in Pediatric Patients With Tourette Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tasly Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: T92-US-01
Record Dates: First submitted 2021-12-23; First posted 2022-01-12 (Actual); Last update posted 2022-01-12 (Actual); Status verified 2022-01

CONDITIONS: Tourette Syndrome in Children; Tourette Syndrome in Adolescence
Keywords: Tourette Syndrome
MeSH Terms: conditions — Tourette Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- T92 group (Experimental): The dose of T92 was calculated based on body weight, orally twice daily. Supportive care duration: 8 weeks
  Interventions: Dietary Supplement: T92
- Placebo group (Placebo Comparator): The dose of placebo was calculated based on body weight, orally twice daily. Supportive care duration: 8 weeks
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: T92 — T92 granules (5g/sachet) will be taken BID for 8 weeks, the dosage will be calculated by individual's body weight.
  Arms: T92 group
Dietary Supplement: Placebo — The placebo matched to T92 granules will be taken BID for 8 weeks.
  Arms: Placebo group

SUMMARY:
A 12-week clinical study to evaluate the safety and efficacy of T92 in pediatric patients with Tourette Syndrome.

DETAILED DESCRIPTION:
This is a multi-center, randomized, double-blind, placebo-controlled, outpatient clinical study designed to evaluate the efficacy and safety of T92 in Tourette Syndrome pediatric patients.

This trial consists of a screening/wash-out period of up to 6 weeks, an 8-week supportive care period and a 4-week follow-up period for all subjects who completed the study. For the first two weeks, the patients will continue to take T92 at half dose and the T92 administration will be stopped from week 3 of the follow-up period.

Subjects will be randomly assigned to receive T92 or matching placebo based on individual body weight. The calculated amount of investigational product (T92 or placebo) will be administrated orally twice daily. Morning dose and evening dose should be administrated at about the same time every day and irrelevant to meals.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female children and adolescents aged 6 to 17 years upon screening with a Diagnosis of Tourette Syndrome according to Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-V).
2. TTS ≥ 20 on the YGTSS at screening and baseline.
3. In the Investigator's opinion the presenting tic symptoms caused impairment in the subject's normal daily routines.
4. Females of childbearing potential had a negative pregnancy test, practiced acceptable double-barrier methods of contraception (or abstinence), and were not pregnant or lactating.
5. Written informed assent or consent provided by the subject, and written informed consent provided by the parent(s)/guardians(s), as appropriate per the IRB/EC.
6. In the opinion of the Investigator, the subject and designated guardian(s) and/or parent(s) must be considered likely to comply with the study protocol and to have a high probability of completing the study.

Exclusion Criteria:

1. Medical history consistent with another neurologic condition that may have had accompanying abnormal movements (e.g., Huntington's disease, Parkinson's disease, Sydenham's chorea, Wilson's disease, Mental retardation, Traumatic brain injury, Stroke, Restless legs syndrome)
2. History of schizophrenia, bipolar disorder, or other psychotic disorder; Comorbid conditions such as: Obsessive Compulsive Disorder (OCD) and Attention Deficit Hyperactivity Disorder (ADHD) can be included.
3. Active major depression disorder.
4. History of neuroleptic malignant syndrome.
5. Subjects who have had treatment with:

   1. investigational medication within 3 months of starting study
   2. depot antipsychotics within 3 months of starting study
   3. Antipsychotics with possible effects on TS symptoms: i.e., topiramate within 1 week; levodopa or dopamine agonists within 2 weeks prior to baseline.
   4. VMAT2 inhibitors within 2 weeks prior to baseline.
   5. Atypical antipsychotics within 4 weeks: this class include risperidone (Risperdal), quetiapine (Seroquel), olanzapine (Zyprexa), ziprasidone (Zeldox), paliperidone (Invega), aripiprazole (Abilify) and clozapine (Clozaril).
   6. Selective serotonin reuptake inhibitors unless the dosage has been stable for a minimum of 4 weeks prior to study start and not prescribed to relieve the neurological signs of TS.
6. Sexually active males or females who would not commit to utilizing 2 of the approved birth control methods or who would not remain abstinent during the trial and for 90 days (males) or 30 days (females) following the last dose of investigational product.
7. CBIT need to be started at least two months at screening. Could continue on existing therapy or stop it based on PI's opinion.
8. Significant psychoactive substance use disorder within the past 3 months; or the urine drug screen was positive.
9. Significant lab abnormality:

   1. Platelets ≤ 75,000/mm3
   2. Hemoglobin ≤ 9 g/dl
   3. Neutrophils, absolute ≤ 1000/mm3
   4. Aspartate transaminase (AST) > 3×ULN (upper limit of normal)
   5. Alanine aminotransferase (ALT) > 3×ULN
   6. Creatinine ≥ 2 mg/dl
10. History or presence of any clinically important medical condition that, in the judgment of the investigator, is likely to deteriorate, could be detrimental to the subject, or could affect the subject's ability to complete the study.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Estimated)
Dates: Start 2022-05 (Estimated); Primary Completion 2024-02 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
The mean change from baseline to week 8 in total tic score (TTS) of Yale Global Tic Severity Scale (YGTSS). | Baseline, Week 8
  The Yale Global Tic Severity Scale (YGTSS) is a semi-structured clinical interview for assessing the severity of tics in children and adults. The YGTSS enables evaluations of number, frequency, intensity, complexity, and interference of motor and phonic tics, covering the past week. Each domain is scored on a 6-point scale (range 0-5) with a separate rating for "overall impairment" regarding the subject's daily life and activities. YGTSS-TTS is the sum of the total motor tic score plus the total phonic tic score ranging from 0-50. Higher scores indicate greater severity/worse outcome. Changes in TTS after 8 weeks of supportive care duration will be compared between the T92 and placebo groups.

SECONDARY OUTCOMES:
The change from baseline to Week 8 in total Yale Global Tic Severity Scale (YGTSS) scale YGTSS tic-related impairment (TRI) score at week 8 | Baseline, Week 8
  The YGTSS ranking of impairment (YGTSS-TRI), with a maximum of 50 points, is based on the impact of the tic disorder on areas of self-esteem, family life, social acceptance, and school scores. Higher scores indicate greater severity/worse outcome.
Mean change from baseline to TS-CGI severity and improvement at week 8 | Baseline, Week 2, 4, 6 and 8
  The TS-CGI scale is a 7-point Likert scale that allows the clinician to use all available information to assess the impact of tics on the participant's quality of life. Lower scores indicate better quality of life. Mean score was calculated with T92 and placebo group, on week 2, 4, 6, and 8.
Clinical response rate, defined as a ≥ 30% reduction from baseline on TTS score at different check points. | Baseline, Week 2, 4, 6 and 8
  Clinical response defined as a ≥ 30% reduction from baseline on TTS at week 2, 4, 6 and 8. The clinical response rate is the proportion of subjects who achieve clinical response.
Evaluation of T92 in reducing severity of the sensations before the emergence of tics by comparing the change in PUTS scores at week 8 from baseline. | Baseline, Week 4 and 8
  The PUTS is a nine-item self-reported scale that measures the sensations before the emergence of tics, and each item is scored from 1 to 4. The total score (range: 9-36) is obtained by summing all of the nine items. Higher scores indicate greater severity/worse symptoms.
Evaluation of T92 in reducing severity of obsessions and compulsion occurring by comparing the change in CY-BOCS scores at week 8 from baseline. | Baseline, Week 4 and 8
  The CY-BOCS is assessing the severity of obsessions and compulsion occurring over the past week. OCD severity score (range 0-40) including all 10 items rated on a 5-point Likert scale (range 0-4). Higher scores indicate greater severity/worse symptoms.
Evaluation of T92 in reducing severity of ADHD symptoms. | Baseline, Week 4 and 8
  The ADHD-RS-IV is an 18-item scale based on the DSM-IV-TR criteria for ADHD that provides a rating of the severity of symptoms. The first 9 items assess inattentive symptoms and the last 9 items assess hyperactive-impulsive symptoms. Scoring is based on a 4-point Likert-type severity scale: 0 = none, 1 = mild, 2 = moderate, 3 = severe. Higher scores indicate greater severity/worse symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Michael H Bloch, MD, PhD, Principal Investigator — Yale University
Locations (1):
- Yale Child Study Center, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No